CLINICAL TRIAL: NCT05508542
Title: The Effect of Progressive Relaxation Exercises on Sleep Quality, Anxiety and Stress Levels in Risky Pregnants
Brief Title: Progressive Relaxation Exercises and Sleep, Anxiety and Stress in Risky Pregnants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra ÇERÇER, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Health Care Seeking Behavior
Keywords: risky pregnancy; progressive relaxation exercises; anxiety; stress; nursing
MeSH Terms: conditions — Patient Acceptance of Health Care; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Progressive relaxation exercises (Experimental): Afterwards, the researcher will first give training on progressive relaxation exercises to the patient in the patient's room. A relaxation exercise program will be installed on the patients' phones via the Whatsapp application. It is planned that the trainings will be applied to the patients one-to-one and will last an average of 40-45 minutes for each patient.
  After these trainings are completed, a booklet will be given to the patients that will contribute to the correct practice of relaxation exercises on their own. Patients will be asked to practice relaxation exercises by listening to the programs downloaded to their phones at least three times a week for 4 weeks.
  In the final test phase; Pittsburgh Sleep Quality Index (PUKI), Prenatal Anxiety Screening Scale and Pregnancy Stress Rating Scale will be re-administered 4 weeks after the start of exercise practices.
  Interventions: Behavioral: Progressive relaxation exercises
- No Intervention: Standard care group (No Intervention): Standard care group.

INTERVENTIONS:
Behavioral: Progressive relaxation exercises — Personal information form, Pittsburgh Sleep Quality Index (PUKI), Prenatal Anxiety Screening Scale and Pregnancy Stress Rating Scale will be applied to the pregnant women at the first interview. Afterwards, the researcher will first give training on progressive relaxation exercises to the patient in the patient's room. Afterwards, the Relaxation Exercises CD will be played and the exercises will be performed with the patient along with the CD. A relaxation exercise program will be installed on the patients' phones via the Whatsapp application. It is planned that the trainings will be applied to the patients one-to-one and will last an average of 40-45 minutes for each patient.
  Arms: Intervention group: Progressive relaxation exercises

SUMMARY:
This study was planned as a randomized controlled quasi-experimental study to determine the effect of progressive relaxation exercises on sleep quality, anxiety and stress levels in risky pregnant women. "Personal Information Form", "Pittsburgh Sleep Quality Index (PUKI)" to measure the sleep quality of pregnant women, "Perinatal Anxiety Screening Scale" to determine the anxiety levels of pregnants, "Pregnancy Stress Scale" to determine the perceived stress level of pregnants, which were created by the researchers in the direction of the literature in data collection. Evaluation Scale".The universe of the research, T.C. It will consist of pregnant women who are hospitalized with the diagnosis of risky pregnancy in the Ministry of Health Adana City Training and Research Hospital Gynecology and Obstetrics Clinics. The sample size was determined as 15 patients to compare the means between the two groups. With an expected dropout rate of 10% and to ensure the adequacy of the final sample size, 17 patients were selected per group.Relaxation exercises are easy to apply, economical, safe and effective non-pharmacological applications that can be used independently by nurses and midwives. By ensuring the management of risky pregnancies, it will support the protection and development of public health by ensuring the protection of both women and fetus health.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled quasi-experimental study to determine the effect of progressive relaxation exercises on sleep quality, anxiety and stress levels in risky pregnant women.

H1-1: There is a significant difference between the sleep quality posttest total score averages.

H1-2: There is a significant difference between the anxiety level posttest total score averages.

H1-3: There is a significant difference between the stress level posttest total score averages.

The universe of the research, T.C. It will consist of pregnant women who are hospitalized with the diagnosis of risky pregnancy in the Ministry of Health Adana City Training and Research Hospital Gynecology and Obstetrics Clinics. "Personal Information Form", "Pittsburgh Sleep Quality Index (PUKI)" to measure the sleep quality of pregnant women, "Perinatal Anxiety Screening Scale" to determine the anxiety levels of pregnants, "Pregnancy Stress Scale" to determine the perceived stress level of pregnants, which were created by the researchers in the direction of the literature in data collection. Evaluation Scale".Intervention Group The pregnant women who were diagnosed with a risky pregnancy, admitted to the clinic and met the research participation criteria will be informed about the study by the researchers, and verbal and written consents of the pregnant women who accepted to participate in the study will be obtained and the study will begin.

Personal information form, Pittsburgh Sleep Quality Index (PUKI), Prenatal Anxiety Screening Scale and Pregnancy Stress Rating Scale will be applied to the pregnant women at the first interview. Afterwards, the researcher will first give training on progressive relaxation exercises to the patient in the patient's room. Afterwards, the Relaxation Exercises CD will be played and the exercises will be performed with the patient along with the CD. A relaxation exercise program will be installed on the patients' phones via the Whatsapp application. It is planned that the trainings will be applied to the patients one-to-one and will last an average of 40-45 minutes for each patient.

After these trainings are completed, a booklet will be given to the patients that will contribute to the correct practice of relaxation exercises on their own. Patients will be asked to practice relaxation exercises by listening to the programs downloaded to their phones at least three times a week for 4 weeks. Researchers will follow the patients over the phone for 4 weeks.

In the final test phase; Pittsburgh Sleep Quality Index (PUKI), Prenatal Anxiety Screening Scale and Pregnancy Stress Rating Scale will be re-administered 4 weeks after the start of exercise practices.

Control Group In the control group, pregnant women who meet the research participation criteria will be informed about the study by the researchers, verbal and written consents of the pregnant women who accepted to participate in the study will be obtained and data collection will begin.

The control group will receive routine nursing care in the clinic and no intervention will be made to this group. Pittsburgh Sleep Quality Index (PUKI), Prenatal Anxiety Screening Scale and Pregnancy Stress Rating Scale will be applied at the first interview.

In the post-test phase, 4 weeks after the start of the first interview, the Pittsburgh Sleep Quality Index (PUKI), Prenatal Anxiety Screening Scale and Pregnancy Stress Rating Scale will be administered again.

In order to prevent the pregnant women in the control group from being affected by the pregnant women in the intervention group, pregnant women in different rooms will be selected for the intervention and control group.Progressive relaxation exercises are a non-pharmacological method that can be easily applied by both nurses and pregnant women in the management of life-threatening risky pregnancies for maternal and fetal health. Improving the sleep quality of pregnant women, reducing perceived stress and anxiety levels will increase their quality of life. By ensuring the management of risky pregnancies, it will support the protection and development of public health by ensuring the protection of both women and fetus health. The work done in this area is limited. At the end of the study, it is thought that it will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate,
* No communication problem,
* Not having any psychiatric disease,
* Diagnosed with a risky pregnancy for at least one month,
* In the last trimester of pregnancy,
* Having a smart phone,
* Internet access

Exclusion Criteria:

* Pregnant women diagnosed with restless legs syndrome during treatment and follow-up,
* Women who gave birth before the end of the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — female
Enrollment: 30 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PUKI) | change in sleep quality at four weeks
  It was developed by Buysse et al. in 1989 (Buysse et al., 1989). The Turkish validity and reliability study of the scale was conducted by Ağargün et al. (1996) and the Cronbach Alpha internal consistency coefficient was found to be 0.80.A total score higher than 5 indicates poor sleep quality .

SECONDARY OUTCOMES:
Prenatal Anxiety Screening Scale | change in anxiety level at four weeks
  It was developed by Somerville et al. in 2013 and validated and reliable in 2019 by Yazıcı et al. The scale consists of 31 items. The four sub-dimensions of the scale are: (1) acute anxiety and adjustment disorder, (2) general anxiety and specific fears, (3) perfectionism, control and trauma, and (4) social anxiety. Cronbach Alpha was found to be 0.95. The cut-off point on the original scale was calculated as 26, minimum anxiety symptoms 0-20, mild-moderate 21-41, and severe anxiety 42-93

OTHER OUTCOMES:
Pregnancy Stress Rating Scale (GSDS-36) | change in stress level at four weeks
  The Turkish validity and reliability of the Pregnancy Stress Rating Scale-36 developed by Chung-Hey Chen (2015) was performed by Akın in 2018. It is interpreted that the higher the total score obtained from the scale, the higher the stress. In the validity and reliability study of the scale, the Cronbach Alpa value of GSDS-36 was found to be 0.92

CONTACTS AND LOCATIONS:
Overall Officials: Zehra ÇERÇER, PhD, Principal Investigator — Cukurova University; Evşen NAZİK, Prof. Dr., Study Director — Cukurova University
Locations (1):
- Cukurova Unıversity, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Somerville S, Dedman K, Hagan R, Oxnam E, Wettinger M, Byrne S, Coo S, Doherty D, Page AC. The Perinatal Anxiety Screening Scale: development and preliminary validation. Arch Womens Ment Health. 2014 Oct;17(5):443-54. doi: 10.1007/s00737-014-0425-8. Epub 2014 Apr 4. PMID 24699796
- [Background] Akmese ZB, Oran NT. Effects of Progressive Muscle Relaxation Exercises Accompanied by Music on Low Back Pain and Quality of Life During Pregnancy. J Midwifery Womens Health. 2014 Sep-Oct;59(5):503-9. doi: 10.1111/jmwh.12176. Epub 2014 Jun 25. PMID 24965313